CLINICAL TRIAL: NCT02710942
Title: Testing the Feasibility of Two Self-guided Web-based Interventions for Adolescents and Young Adults With Migraine: A Pilot Randomized Controlled Trial
Brief Title: Testing myWHI: Online Self-guided Programs for Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Anna Huguet, Research Scientist, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSO-EST-2014-9575
Record Dates: First submitted 2015-11-12; First posted 2016-03-17 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SPHERE intervention (Experimental): It is a comprehensive self-guided Internet-based cognitive-behavioral therapy (CBT) that includes three components: (1) the myWHI diary. (2) 30 multi-media learning topics that the user is encouraged to go through in a sequential way. The topics contain education information and teach strategies to cope better with their headaches.
  Interventions: Behavioral: SPHERE
- PRISM intervention (Experimental): It is a targeted self-guided Internet-based CBT intervention. PRISM was built upon the myWHI diary, an electronic headache diary. PRISM helps users discover their headache triggers by analyzing the inputted diary data using association rule mining. Once one or multiple headache triggers are identified the application uses an algorithm to provide the user with a few personalized recommendations to help them to cope with these triggers. The algorithm is based on the opinion of clinical experts (e.g., medical health professionals, psychologists). The user chooses recommendations to follow and sets goals in the application to follow them. To support the process, the application checks in with users about their goals and tracks goal completion.
  Interventions: Behavioral: PRISM
- Usual care (No Intervention): Participants can continue doing what they usually do to deal with their migraines.

INTERVENTIONS:
Behavioral: SPHERE
  Arms: SPHERE intervention
Behavioral: PRISM
  Arms: PRISM intervention

SUMMARY:
The goal for this pilot study is to assess the acceptability of two online self-guided programs for migraines. The programs are part of the investigators' collection of "my Wireless Headache Interventions" (myWHI). The Specialized Program for Headache Reduction (SPHERE) is a program that teaches cognitive and behavioural skills/techniques to help manage headaches. The PeRsonalized Intervention for Self-Management of Migraine (PRISM) helps users to discover their headache triggers and provides recommendations for managing them. This pilot will also assess the feasibility of the study protocol to inform a full scale randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* aged 14-35 years
* fluent in the English language (i.e., speaking, reading and writing);
* suffer from headaches for a minimum of one year
* stable pattern of headache symptoms (e.g., headache frequency, severity, location of pain, symptoms associated with headache) for the past 6 months
* suffer from migraine headaches as indicated with a score of 2 and above on the ID Migraine
* use the Smartphone for activities other than texting and calling (e.g., email, Facebook)
* have daily Internet access from their Smartphone
* minimum of four headache days during 4 weeks of using an electronic headache diary

Exclusion Criteria:

* health care professional has not ruled out any underlying medical condition related to their headaches (e.g., head trauma, meningitis)
* are pregnant, planning to get pregnant (in the next 4 to 6 months), or breastfeeding
* have an impairment which compromises their ability to give informed consent
* having been diagnosed with psychosis and/or schizophrenia
* they complete less than 50% of daily entries (i.e., less than 14 daily entries) in an electronic headache dairy

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Average number of individuals who complete the online screening per month | After reaching our desired sample size for randomization
  This is an exploratory study and we do not know how much time it will take for us to recruit our desired sample size. However, our maximum time frame is 1 year.
Proportion of recruited participants who are eligible for study entry | After reaching our desired sample size for randomization
  This is an exploratory study and we do not know how much time it will take for us to recruit our desired sample size. However, our maximum time frame is 1 year.
Proportion of eligible participants who consent | After reaching our desired sample size for randomization
  This is an exploratory study and we do not know how much time it will take for us to recruit our desired sample size. However, our maximum time frame is 1 year.
Proportion of consented participants who are randomized | After reaching our desired sample size for randomization
  This is an exploratory study and we do not know how much time it will take for us to recruit our desired sample size. However, our maximum time frame is 1 year.
Proportion of randomized participants who drop out | At 4-month post-randomization
Level of usage of the Internet-based interventions (i.e., PRISM and SPHERE). Intervention usage will be tracked automatically | At 4-month post-randomization
Proportion of consented participants who complete the baseline assessment | After reaching our desired sample size for randomization
  This is an exploratory study and we do not know how much time it will take for us to recruit our desired sample size. However, our maximum time frame is 1 year.
Proportion of randomized participants who complete the 4-month post-randomization assessment | At 4-month post-randomization
Acceptability of the Internet-based interventions (i.e., PRISM and SPHERE) using the 8-item Client Satisfaction Questionnaire (CSQ-8) | At 4-mont post-randomization
Acceptability of the Internet-based interventions (i.e., PRISM and SPHERE) using the single-item Patients' Global Impression of Change Scale (PGIC) | At 4-mont post-randomization
Acceptability of the Internet-based interventions (i.e., PRISM and SPHERE) using the satisfaction interviews | At 4-mont post-randomization
Proportion of participants in the control group who show clinically significant improvement (50% or greater reduction) from baseline in number of headache days in the last 4 weeks | At 4-mont post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Anna Huguet, PhD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No